CLINICAL TRIAL: NCT02911155
Title: Cancer and Other Disease Risks in U.S. Nuclear Medicine Technologists
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916141; 16-C-N141
Record Dates: First submitted 2016-09-21; First posted 2016-09-22 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Brain Cancer; Thyroid Cancer; Circulatory Disease; Breast Cancer
Keywords: Cohort Study; Radiation; Occupation
MeSH Terms: conditions — Brain Neoplasms; Thyroid Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- US Nuclear Medicine Technologist: radiologic technologists certified in nuclear medicine

SUMMARY:
Background:

The field of nuclear medicine has changed a lot in the past decades. Technology has gotten better, so patients are exposed to less radiation. But now workers are doing procedures more often and using lead aprons less. So they may be exposed to more radiation. This may put them at higher risk for cancers and other health problems that are related to radiation. Researchers want to collect data from technologists to learn more about the risks and appropriate doses of radiation.

Objective:

To learn more about the risks and appropriate doses of radiation for nuclear medicine technologists.

Eligibility:

Adults who were first certified in nuclear medicine technology in the United States after 1980. They must be living in the United States. They must not be participants in the USRT study.

Design:

Participants will be recruited online.

Participants will complete an online survey. It will take about a half hour. This will have questions about their work with nuclear medicine procedures. There will be questions about the kinds of procedures and how often they do them.

Participants will give a short work history. This will include the names of current and past employers.

Participants will allow researchers to get records of their film badge dose readings. These will come from dosimetry providers.

Dosimetry data will not be shared with participants. Researchers can t ensure the how accurate or complete the data are.

DETAILED DESCRIPTION:
The field of nuclear medicine has expanded rapidly since its inception in the mid-20th century, with nuclear medicine technologists now potentially experiencing higher levels of radiation exposure relative to other medical worker populations. Many radiopharmaceuticals and procedures used in previous decades are now obsolete and are being replaced by new and emerging radioisotopes and combined-modality and molecular imaging procedures. While improvements in imaging technologies and the introduction of certain radioisotopes have generally reduced patient exposure to radiation, nuclear medicine technologists have become increasingly specialized in these newer procedures and are performing these and other nuclear medicine procedures with increasing frequency. Furthermore, lead aprons are less effective in protecting workers during nuclear medicine procedures, specifically higher-energy procedures (e.g., positron emission tomography (PET)), compared to other radiation-related procedures, and are seldom used by technologists performing nuclear medicine. As a result, cumulative doses to nuclear medicine technologists are expected to have increased. We hypothesize that certified nuclear medicine technologists may experience higher risks of some radiation-related cancers and other adverse health outcomes compared to most other medical specialty groups. There is currently very little information about radiation-related risks associated with performing these procedures due, in part, to limited information on occupational doses associated with current nuclear medicine practices. To characterize organ-specific doses that could later be used to quantify risks for specific radiation-related disease outcomes, either directly (through subsequent follow-up) or indirectly (through risk projection methods), we plan to collect detailed work history information on nuclear medicine procedures and associated radiation safety practices, as well as badge doses, for a representative sample of 1,500 technologists certified in nuclear medicine in the U.S. This information will complement similar data collected in 2013-2014 from an independent sample of approximately 4,500 general radiologic technologists in the U.S. Radiologic Technologists Study (USRT) who had reported working with these procedures. However, unlike the USRT sample, the proposed sample is expected to be higher-risk, including only those workers with a specialty certification in nuclear medicine who will have been begun working with nuclear medicine procedures much earlier in their career, at ages associated with greater susceptibility to radiation-related carcinogenesis.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Technologists from the target population of approximately 25,000 individuals who were first certified in nuclear medicine technology in the U.S. after 1980, are currently alive and residing in the U.S., and are not participants of the USRT study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an occupational cohort of 35,593 U.S. nuclear medicine technologists certified by the American Registry of Radiologic Technologist or the Nuclear Medicine Technology Certification Board in 1980 or later.
Sampling Method: Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2016-09-21; Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
U.S. nuclear medicine tecnologist | 2016-2022
  Cancer and other disease risks associated with occupational nuclear medicine radiation exposures

SECONDARY OUTCOMES:
Administer questionnaire | 2016-2018
  Collect data on nuclear medicine procedures performed, radioisotopes used, related work and safety practices, and places of employment over time.
Obtain badge doses | 2016-2019
  Collect badge doses from the nation's largest commercial dosimetry provider for use in estimating occupational radiation exposures.

CONTACTS AND LOCATIONS:
Overall Officials: Cari M Kitahara, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Minnesota, School of Public Health Environmental Health Sciences, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Drozdovitch V, Brill AB, Callahan RJ, Clanton JA, DePietro A, Goldsmith SJ, Greenspan BS, Gross MD, Hays MT, Moore SC, Ponto JA, Shreeve WW, Melo DR, Linet MS, Simon SL. Use of radiopharmaceuticals in diagnostic nuclear medicine in the United States: 1960-2010. Health Phys. 2015 May;108(5):520-37. doi: 10.1097/HP.0000000000000261. PMID 25811150
- [Background] Kitahara CM, Linet MS, Drozdovitch V, Alexander BH, Preston DL, Simon SL, Freedman DM, Brill AB, Miller JS, Little MP, Rajaraman P, Doody MM. Cancer and circulatory disease risks in US radiologic technologists associated with performing procedures involving radionuclides. Occup Environ Med. 2015 Nov;72(11):770-6. doi: 10.1136/oemed-2015-102834. Epub 2015 Jul 28. PMID 26220810
- [Background] Drozdovitch V, Brill AB, Mettler FA Jr, Beckner WM, Goldsmith SJ, Gross MD, Hays MT, Kirchner PT, Langan JK, Reba RC, Smith GT, Bouville A, Linet MS, Melo DR, Lee C, Simon SL. Nuclear medicine practices in the 1950s through the mid-1970s and occupational radiation doses to technologists from diagnostic radioisotope procedures. Health Phys. 2014 Oct;107(4):300-10. doi: 10.1097/HP.0000000000000107. PMID 25162420